CLINICAL TRIAL: NCT07371299
Title: Multimodal Objective Measures Help Cochlear Implant Programming: Cross-sectional and Prospective Study Focusing on the Correlations Between eSRT, Behavioural and Other Objective Responses (eABR, eCAP)
Brief Title: Correlations Between Subjective and Objective Responses to Cochlear Implant Stimulation
Acronym: CRSOSIC
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Cochlear (Industry)
Responsible Party: Sponsor
Other Study IDs: APHP250486; 2025-A01446-43 (Other: IDRCB)
Record Dates: First submitted 2025-11-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Severe to Profound Sensorineural Hearing Loss
Keywords: Cochlear implants; Cochlear implant stimulation; Electrical compound action potentials (eCAP); Electrical auditory brainstem response (eABR); electrical stapedius reflex threshold (eSRT)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Incident CI Cohort (Prospective Adults): Adults ≥18 scheduled for first-time unilateral cochlear implantation within 3 months; followed post-op at M1, M3, M6, M9, M12. Objective measures on ≥3 electrodes (basal, middle, apical): eCAP via CI software; eABR via evoked-potential system; eSRT via tympanometer. No experimental intervention (routine programming only). Main interest: associations between objective metrics and behavioral MCL, with key analyses at M6 and M12.
  Interventions: Diagnostic Test: Objective electrophysiological measures (eCAP, eABR, eSRT)
- Prevalent CI Cohort (Cross-Sectional Adults): Adults ≥18 with unilateral cochlear implant use ≥12 months; single annual follow-up visit. Same objective measures (eCAP, eABR, eSRT) on ≥3 electrodes using standard clinical equipment; no intervention. Purpose: cross-sectional correlations and comparison with the incident cohort.
  Interventions: Diagnostic Test: Objective electrophysiological measures (eCAP, eABR, eSRT)

INTERVENTIONS:
Diagnostic Test: Objective electrophysiological measures (eCAP, eABR, eSRT) — Non-invasive electrophysiological recordings obtained during/after routine cochlear-implant programming, using standard clinical equipment: eCAP via CI software, eABR via an evoked-potential system synchronized with the implant, and eSRT via tympanometry. No investigational device or randomization. Measurements are collected for observational correlations with behavioral levels. Schedule: incident cohort at M1, M3, M6, M9, M12; prevalent cohort single annual visit.

SUMMARY:
Cochlear implants have been used for several decades, with major technological advances. However, adjustment can be difficult for patients who have to get used to a new sound that is electrical rather than acoustic. In general, adjustment is based on the patient's responses: the patient must inform the technician of their sensations in order to determine the sound level that is comfortable for them (MCL: maximum comfortable level).

The adjustment therefore depends on a subjective assessment. The aim of the adjustments is to make the sound pleasant while increasing the stimulation level to the maximum tolerated level in order to achieve good listening dynamics. Objective indicators would therefore be useful in improving the accuracy of the adjustments. The objective measurements that can be taken are:

* Electrical compound action potentials (eCAP)
* Electrical auditory brainstem response (eABR)
* Electrical stapedius reflex threshold (eSRT).

DETAILED DESCRIPTION:
Observational study of adult patients who are going to receive or have received a cochlear implant. In fact, two groups of patients will be studied:

Incident case cohort: patients included in the cohort will be followed for one year after surgery.

Data will be collected at each postoperative follow-up visit (M1, M3, M6, M9, M12) to monitor their progress. Each objective measurement will be taken on at least three electrodes: on the left, right, and central electrodes. Data will be collected at each postoperative follow-up visit (M1, M3, M6, M9, M12) in order to monitor their progress. Each objective measurement will be taken on at least three electrodes: on the basal, median, and apical parts of the electrode array. Stimulation will be configured using the software normally used to adjust the implant.

Responses are collected:

* for eCAPs: via the same software
* for eABRs: using an auditory evoked potential recording device synchronized with the implant stimulations
* for eSRTs: using a tympanometer with the probe inserted into the external auditory canal on the same side or the opposite side to the stimulation. Cross-sectional sample of prevalent cases: The same measurements will be taken in patients who had a cochlear implant some time ago (evaluation more than one year after surgery). The measurements will be taken only once during their annual check-up. This population will enable us to compare data from patients who have recently had an implant with data from a population that already has a minimum of experience and adaptation to the implant.

ELIGIBILITY:
Inclusion Criteria:

Incident case cohort:

* Age ≥ 18 years (18 years or older)
* Scheduled for first-time unilateral cochlear implantation within the next 3 months
* Informed about the study and did not object (non-opposition)

Cross-sectional sample of prevalent cases:

* Age ≥ 18 years (18 years or older)
* Underwent unilateral cochlear implantation more than 1 year ago
* Has used the implant for more than 1 year (interval between implantation surgery and study inclusion > 1 year)
* Informed about the study and did not object (non-opposition)

Exclusion Criteria:

Exclusion Criteria - applies to both the incident case cohort and the cross-sectional sample of prevalent cases:

* Prior middle or inner ear surgery
* Cognitive impairment or insufficient comprehension of French that would prevent understanding of study procedures or accurate measurement of comfort thresholds during programming
* Peripheral facial palsy
* Bilateral cochlear implantation
* Patient under legal guardianship/court-ordered protection

Additional exclusion - cross-sectional sample of prevalent cases only:

- More than half of the electrodes not inserted (i.e., <50% electrode insertion)

Secondary exclusion criteria - Incident case cohort:

* More than half of the electrodes not inserted (<50% electrode insertion)
* Postoperative peripheral facial nerve palsy following the implantation surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are going to receive or have received a cochlear implant.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
The MCL threshold, the objective response threshold (eSRT), the eSRT response | 15 months
  "The MCL threshold, expressed in CU (charge unit) units, corresponds to the maximum level of stimulation of the implant required to obtain a sound level considered comfortable by the patient. It will be recorded at each post-operative check-up (M1, M3, M6, M9, and M12).
  The objective response threshold (eSRT), expressed in CU units, corresponds to the minimum level of implant stimulation required to elicit a stapedial reflex. It will be recorded at each post-operative assessment (M1, M3, M6, M9, and M12).
  The eSRT response will be collected using a tympanometry probe (commonly used to measure ear impedance in patients during a standard hearing assessment) in the patient's external auditory canal, ipsilateral or contralateral to the implanted side. The tympanometer will continuously record ear impedance during electrical stimulation until a significant variation is obtained, indicating the presence of the stapedial reflex."

SECONDARY OUTCOMES:
Correlation between behavioral MCL and eABR threshold | Month 6 and Month 12 post-operative follow-up visits (incident cohort)
  Pearson/Spearman correlation between Maximum Comfortable Level (MCL, charge units [CU]) and electrically evoked Auditory Brainstem Response (eABR) threshold (CU); measured on ≥3 electrodes (basal, middle, apical) using standard CI programming and evoked-potential equipment.
Correlation between behavioral MCL and eCAP threshold | M1, M3, M6, M9, M12 post-operative visits (incident cohort).
  Pearson/Spearman correlation between MCL (CU) and electrically evoked Compound Action Potential (eCAP) threshold (CU); measured on ≥3 electrodes (basal, middle, apical) via implant software.
Correlation between eSRT and eABR thresholds | M6 and M12 post-operative visits (incident cohort).
  Pearson/Spearman correlation between electrically evoked Stapedius Reflex Threshold (eSRT, CU) and eABR threshold (CU); ≥3 electrodes per visit.
Correlation between eSRT and eCAP thresholds | M1, M3, M6, M9, M12 post-operative visits (incident cohort).
  Pearson/Spearman correlation between eSRT (CU) and eCAP threshold (CU); ≥3 electrodes per visit.
Correlation between eABR and eCAP thresholds | Month 6 and Month 12 after cochlear implantation (incident cohort)
  Pearson/Spearman correlation between eABR and eCAP thresholds (both in CU); ≥3 electrodes per visit.
Agreement between intraoperative eSRT by tympanometer vs visual stapedius reflex | ntraoperative (single time point during CI surgery).
  Association between peri-operative eSRT measured objectively with a tympanometer and the surgeon's visual observation of stapedius movement (yes/no).
Probe frequencies eliciting eSRT | Post-operative follow-up visits at Month 1, Month 3, Month 6, Month 9, and Month 12 (incident cohort), and 1 year or more after cochlear implantation (prevalent cohort)
  Distribution of probe frequencies (226, 678, 1000 Hz) that yield an eSRT response; eSRT level recorded for each tested frequency.
Longitudinal profile of objective thresholds (eSRT/eABR/eCAP) | From Month 1 to Month 12 after cochlear implantation (incident cohort)
  Trajectory of eSRT, eABR, and eCAP thresholds over the first post-operative year, summarized graphically and descriptively.
Cross-sectional associations among MCL and objective measures in prevalent users | At the annual follow-up visit, at least 12 months after cochlear implant surgery.
  Correlations between MCL and eSRT/eABR/eCAP, and pairwise correlations among objective measures, in adults with ≥12 months of CI use.
Between-cohort comparison of correlation coefficients (prevalent vs incident) Description: Comparison of correlation coefficients for each pair (MCL-eSRT, MCL-eABR, MCL-eCAP, eSRT-eABR, eSRT-eCAP, eABR-eCAP) between the prevalent cross-section and the in | Incident cohort: post-operative follow-up visits from Month 1 through Month 12. Prevalent cohort: annual follow-up visit, at least 12 months after cochlear implant surgery.
  Between-cohort comparison of correlation coefficients (prevalent vs incident) Description: Comparison of correlation coefficients for each pair (MCL-eSRT, MCL-eABR, MCL-eCAP, eSRT-eABR, eSRT-eCAP, eABR-eCAP) between the prevalent cross-section and the incident cohort.